CLINICAL TRIAL: NCT04944004
Title: Effectiveness of Computer-based Cognitive Training for Executive Functions After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TWGHs Wong Tai Sin Hospital (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Li Kwok Fai Ray, Mr. Ray Li, TWGHs Wong Tai Sin Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HongKongPolyuRL
Record Dates: First submitted 2021-06-22; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Stroke; Executive Dysfunction; Cognitive Impairment; Randomized Controlled Trial
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental CBCT Group (Experimental): Participants of CBCT group will attend individual computer-based cognitive training sessions. Researcher will give instruction in the use of the computerized training programs and assists participants during their training sessions.
  Interventions: Other: CogniPlus
- Training As Usual (TAU) Group (Active Comparator): Participants of TAU group will attend usual training sessions offered by the training centres with similar intensity and frequency as the CBCT training.
  Interventions: Other: Training As Usual (TAU)

INTERVENTIONS:
Other: CogniPlus — The CBCT programmes proposed in this study is called CogniPlus. This software package offers training of scientifically proven trainable cognitive functions. According to the user manual, the lifelike interactive system and its automatic adaptability to client's ability level made CogniPlus feasible in community settings.
  Arms: Experimental CBCT Group
Other: Training As Usual (TAU) — Training As Usual (TAU)
  Arms: Training As Usual (TAU) Group

SUMMARY:
Objective:

To determine the efficacy of computer-based cognitive training(CBCT) in patients with stroke in the community settings.

Study Design:

Single-blinded prospective, pre-test/post-test randomized controlled trial (RCT) will be conducted in 2 groups of participants that receiving training in community settings. Treatment groups will attend individualized CBCT programme using CogniPlus® while control group will continue attend conventional treatment as usual (TAU). Assessment on the means difference in assessing functions will be done after the study.

Samples:

100 patients with stroke will be recruited from the community, using a sampling frame of selected diagnosis and homogeneity.

Expected Findings:

Find out the training effects of selected CBCT on EF and daily functioning in patients with stroke

DETAILED DESCRIPTION:
It is important to study the effectiveness of intervention post-stroke cognitive deficits in EF, Post-stroke patients with EF deficits will affect their abilities to successfully return to normal daily activity. Studies over the past decade have provided evidence of substantial gaps in our knowledge on how to effectively manage EF impairment post-stroke. To address these gaps there has been growing attention and research into the management of EF impairment post-stroke. Studies have been conducted to address some of these gaps specific to EF impairment and intervention research, and to investigate use of evidence-based practices for the management of EF impairment post-stroke. The literatures review of EF interventions identified different treatment approaches that were showing promise in helping persons with stroke to cope with EF deficits. The preliminary evidence on specific EF skill retraining suggested that structured, individualized, and intense computerized EF training could improve targeted EF impairments. Stroke patients with EF deficits often find it difficult in their daily activities, the impact of treatment might have potential to enhance rehabilitation and recovery. The translational framework described in (figure IV) describe ways to identify and investigate the evidence for the use of CBCT in specific EF interventions post-stroke. The study is thus required to find the impact of CBCT on a variety of outcomes, including not only measures of EF impairment, but also measures of daily activities and participation in everyday life situations that are affected in stroke patients having EF disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are suffered from unilateral hemispheric stroke and with a confirmation by neuroimaging evidence from either computer tomography (CT) or magnetic resonance imaging (MRI);
2. Patients are either at subacute stage or chronic stage, i.e. the patients are suffered from post-stroke after one month,
3. Patients are age 60 years old or above;
4. Patients are medically stable;
5. Patients are Cantonese speaking,
6. Patients can communicate and to follow at least three-step commands, and;
7. Patients are willing to give written consent.

Exclusion Criteria:

1. Patients are at acute stage, i.e the patients are suffered from stroke within 1 week;
2. Patients with severe aphasia, swallowing disorders or other complications post-stroke that prevent them from successfully completing the assessments;
3. Patients with any previously known psychiatric disorder or neurological disease excluding stroke;
4. Patients are unable to given written consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of Wisconsin Card Sorting Test Score | Baseline, after completion of half of the programme (an average of 8 weeks), one month post-treatment
  The test consists of 128 card designs, participant is required to sort the cards under the categorization rules and feedback from examiner in about 20 minutes. The more categories achieved (range 0 to 6) and less perseverative errors (out of 128 trials) the better executive control. Moreover, the lower the total number of trials administered (total number of cards used) reflects greater efficiency of the participant in the task; in addition, the greater the total number of correct responses (number of successes in combinations according to the category) and the lower the total number of errors (number of incorrect combinations) also indicate the better the participant's performance.

IPD SHARING:
Plan to Share IPD: No